CLINICAL TRIAL: NCT00159055
Title: Prevention and Treatment of CMV Disease by Adoptive Immunotherapy With Immune Donor Lymphocytes in Conjunction With Non-myeloablative Stem Cell Transplantation (NST)
Brief Title: Adoptive Immunotherapy for CMV Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: the PI is no longer work at Hadassah
Sponsor: Hadassah Medical Organization (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 280303-HMO-CTIL
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2011-04-08 (Estimated); Status verified 2005-09

CONDITIONS: CMV Disease
MeSH Terms: interventions — mRNA-1647 cytomegalovirus vaccine

INTERVENTIONS:
Biological: CMV vaccine

SUMMARY:
Treatment strategy of patients:

Stem cell engraftment (myeloablative or NST) for induction of host vs graft myeloablative transplantation tolerance.

Whenever indicated, additional post NST DLI given in graded increment, to optimize control of GVHD.

Preparation of immune donor lymphocytes, either by donor immunization in-vitro with a CMV-specific peptide followed by administration of immunized donor lymphocytes, or by injection of donor lymphocytes and in-vivo sensitization of donor lymphocytes in the patient following DLI.

Pre-emptive treatment of seronegative patients at risk or patients with documented viremia or CMV disease with CMV-specific donor lymphocytes generated in-vivo in the donor or in the host by peptide immunization.

Consenting donors will be immunized with CMV-specific peptides, for induction of CTLs in-vivo following subcutaneous inoculation of peptides with adjuvant or donor APC pulsed with relevant peptides.

ELIGIBILITY:
Inclusion Criteria:

* For Patient:
* Consenting patients with indication for myeloablative BMT or NST with an HLA matching sibling available, for transplant.
* Patients at risk of CMV disease including seronegative patients; patients with seronegative donors, and seronegative donor for sero positive patients.
* Patients with resistant CMV viremia or CMV disease not responding to conventional treatment with ganciclovir, or Foscarnet.
* Patients with HLA phenotype for which a relevant peptide for CMV exists.
* For Donor:
* Consenting sibling >18 years old.
* HLA phenotype for which a relevant peptide for CMV exists.

Exclusion Criteria:

* For Patient:
* Patients with severe resistant GVHD where there may be a risk to administer DLI or immunized donor lymphocytes.
* For Donor:
* Consenting sibling >18 years old.
* HLA phenotype for which a relevant peptide for CMV exists.
* Donor with an infectious disease (e.g. HIV-1; HBV, etc.)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2004-02

PRIMARY OUTCOMES:
Induce and amplify T cell-mediated immunotherapy against cytomegalovirus (CMV) infection in stem cell allograft recipients.

SECONDARY OUTCOMES:
Evaluate toxicity of the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Shimon Slavin, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel